CLINICAL TRIAL: NCT03860506
Title: A Double-Blind, Placebo-Controlled, Randomized, Single-Dose, 2-Period Crossover Study of the Pharmacodynamics of Orally Administered PSI-697 in Healthy Subjects Who Smoke
Brief Title: Study Evaluating the Effects of PSI-697 on Platelets in Subjects Who Smoke
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3165A1-1108; NCT00719069 (obsolete NCT alias)
Record Dates: First submitted 2018-01-22; First posted 2019-03-04 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Healthy
Keywords: healthy subjects who smoke; healthy subjects
MeSH Terms: interventions — 2-(4-chlorobenzyl)-3-hydroxy-7,8,9,10-tetrahydrobenzo(H)quinoline-4-carboxylic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PSI-697 (Experimental)
  Interventions: Drug: PSI-697
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PSI-697
  Arms: PSI-697
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a single dose inpatient and outpatient study to test whether an effect on the ability of platelets to stick to white blood cells in subjects who smoke.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, and 12?lead electrocardiogram (ECG).
* Smoker of at least 1 pack or more of cigarettes per day (20 plus or minus 3 cigarettes) for more than 1 year as determined by history.

Exclusion Criteria:

Exclusion Criteria:

* Any diagnosed bleeding disorder.
* Any major surgical procedure within 6 months before study day 1.
* Any history of major bleeding (eg, bleeding peptic ulcer) within 1 year before study day 1.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-04-01 (Actual); Primary Completion 2008-07-01 (Actual); Study Completion 2008-07-01 (Actual)

PRIMARY OUTCOMES:
reduction of platelet monocyte aggregates | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3165A1-1108&StudyName=Study%20Evaluating%20the%20Effects%20of%20PSI-697%20on%20Platelets%20in%20Subjects%20Who%20Smoke